CLINICAL TRIAL: NCT01699854
Title: Capsaicin Patch 8 % for the Treatment of Persistent Pain After Inguinal Herniotomy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Expiration of the placebo patch
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Joakim Bischoff, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-4-2012-055; 2012-001540-22 (EudraCT Number)
Record Dates: First submitted 2012-09-21; First posted 2012-10-04 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Persistent Pain After Inguinal Herniotomy
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- capsaicin patch (Active Comparator)
  Interventions: Drug: capsaicin patch (qutenza)
- placebo patch (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: capsaicin patch (qutenza)
  Arms: capsaicin patch
Drug: Placebo
  Arms: placebo patch

SUMMARY:
In the present study the investigators intend to investigate analgesic and sensory effects of a capsaicin patch 8 %(Qutenza) in patients with severe post-herniotomy pain and sensory abnormalities in the skin.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA (American Society´s of Anesthesiology´s classification) scores I-III
* Severe post-herniotomy pain for more than six months and with severe pain (numerical rating scale [NRS] 0-10 points) during rest or during movement > 5.

Exclusion Criteria:

* History of an allergic reaction or intolerance to capsaicin or vehicle ingredients in the patches
* Severe cardiac impairment, e.g., NYHA (New York Heart Association) Class ≥ III
* Inflamed or injured skin at the application site
* Signs of cognitive impairment
* Known drug or ethanol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pain change capsaicin vs. placebo patch treatment | Pain intensity assessed at baseline and at 1,2,3 months follow-up
  Summed pain intensity (SPI) is calculated as median pain intensities at rest, during transition from the supine lying to the standing erect position, and auto-palpation twice each day for the last 3 days at baseline and at 1 months, 2 months and 3 months during follow-up. The primary outcome measure is the maximum difference between the summed pain intensity differences (SPID) for the phases: Baseline, 1 month, 2 month or 3 month. Δ SPID is then calculated as the difference in SPID between capsaicin and placebo treated patients.

SECONDARY OUTCOMES:
Changes in AAS (Activities Assessment Scale) score
Changes in HADS (Hospital Anxiety and Depression Scale) score
Changes in QST (Quantitative sensory testing)
Changes in sleep (Sleep Interference Scale) score
Changes in S-LANSS (Leeds self-assessment of neuropathic symptoms and signs)
Changes in intraepidermal nerve fiber density
Subgroup analysis for pain change(summed pain intensity differences (SPID) capsaicin patch vs. placebo are made for patients with thermal hypoesthesia and thermal normo/hyperesthesia
Changes in PCS (Pain Catastrophizing Scale) score

OTHER OUTCOMES:
interim analyses
  An interim analysis evaluating pain change (SPID) for capsaicin patch vs. placebo treatment by an independent statistician following completion of 32 patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen Ø, Denmark

REFERENCES:
- [Derived] Bischoff JM, Ringsted TK, Petersen M, Sommer C, Uceyler N, Werner MU. A capsaicin (8%) patch in the treatment of severe persistent inguinal postherniorrhaphy pain: a randomized, double-blind, placebo-controlled trial. PLoS One. 2014 Oct 7;9(10):e109144. doi: 10.1371/journal.pone.0109144. eCollection 2014. PMID 25290151